CLINICAL TRIAL: NCT01629186
Title: Nasopharyngeal Oxygen With Nose-close and Abdomen-compression in Pediatric Flexible Bronchoscopy
Brief Title: Nose-close and Abdomen-compression in Pediatric Flexible Bronchoscopy
Acronym: NPO-NC-AC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cho-yu Chan, MD (Other Government)
Responsible Party: Sponsor-Investigator, Cho-yu Chan, MD, Taipei Veterans General Hospital,Taiwan, Taipei Veterans General Hospital,Taiwan, Taipei Veterans General Hospital, Taiwan
Organization: Taipei Veterans General Hospital, Taiwan (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VGH-94-269C; NPO-NC-AC in Ped. FB (Other Grant/Funding Number: VGH-94-269C)
Record Dates: First submitted 2011-09-12; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Bradycardia; Hypoxemia
Keywords: CPR; flexible bronchoscope; resuscitation; ventilation
MeSH Terms: conditions — Bradycardia; Hypoxia; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- outcome (Experimental): Cardiopulmonary parameters were measured and recorded at baseline, just before and at every minute during NC-AC, and at the end of the FB session. In infants who already had an arterial line, arterial blood gas (ABG) analyses were taken for study. Data was represented as mean ± SD. The results obtained from the baseline and different stages. The values were considered statistically significant only when p < 0.05.
  Technique failure was defined as: any vital signs of hypoxia did not return to accepted levels(HR>100 beat/min, SpO2>90%, mean BP>50 mmHg)within 2 minutes of the experimental CPR technique. Then traditional CPR procedures involving bag-mask ventilation, endotracheal intubation, Ambu bag ventilation or even chest compressions were substituted.
  Interventions: Other: NPO with Nose-close and Abdomen-compression

INTERVENTIONS:
Other: NPO with Nose-close and Abdomen-compression — Infants with body weight (BW) <5.0 kg and receiving nasal diagnostic or interventional FB were enrolled. Under NPO (0.5 L/kg/min), when infant's heart rate (HR) <80 beats/min or oxygen saturation (SpO2) <85% for more than 10 seconds, rescue NC-AC was initiated. It was performed by (1) increased NPO flow to 0.5-1.0 L/kg/min; (2) NC 1 second for inspiration; and (3) AC 1 second for expiration with simultaneously released nostrils. Repeat doing steps (2) and (3) at a rate of 30 cycles/min until HR, SpO2, and blood pressure (BP) returned to normal.
  Other Names: (1)Nasopharygeal oxygen; (2)Nose-close and Abdomen-compression

SUMMARY:
The nasopharyngeal oxygen (NPO) with Nose-close (NC) and Abdomen-compression (AC) technique may use for support or rescue asphyxiated infants during Flexible bronchoscopy.

DETAILED DESCRIPTION:
OBJECTIVES: To evaluate the efficacy of a novel cardiopulmonary resuscitation (CPR) technique-nasopharyngeal oxygenation with nose-close and abdomen-compression (NPO-NC-AC)-in small infants during flexible bronchoscopy (FB).

METHODS: Infants with body weight (BW) <5.0 kg and receiving nasal diagnostic or interventional FB (dFB, iFB) were enrolled. Under NPO (0.5 L/kg/min), when infant's heart rate (HR) <80 beats/min or oxygen saturation (SpO2) <85% for more than 10 seconds, rescue NC-AC was initiated. It was performed by (1) increased NPO flow to 0.5-1.0 L/kg/min; (2) NC 1 second for inspiration; and (3) AC 1 second for expiration with simultaneously released nostrils. Repeat doing steps (2) and (3) at a rate of 30 cycles/min until HR, SpO2, and blood pressure (BP) returned to normal. Cardiopulmonary parameters were monitored and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* body weight (BW) less than 5.0 kg;
* receiving nasal approach flexible bronchoscopy.

Exclusion Criteria:

* cannot nasal approach flexible bronchoscopy.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 156 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Heart rate (beat/min) | Participants will continually monitoring by EKG for 2 days after the procedure.
  During and after this FB procedure, vital signs are continually monitoring. When the heart rate (HR) <80 beat/min (measured by continuouse wave and digit form of EKG monitor) and lasting >10 seconds. Immediately rescued with rhythmic NC-AC. If the heart rate did not reach to its acceptable level (>80 beat/min) within 2 minutes, then traditional CPR procedures involving bag-mask ventilation, ET intubation, Ambu bag ventilation or even chest compressions were substituted.

SECONDARY OUTCOMES:
Oxygen saturation by pulse oximetry | Participants will continually monitoring by pulse oximeter for 2 days after the procedure.
  During FB procedure, vital signs are continually monitoring. When the oxygen saturation <85% (or more than 10% below the original baseline in already cyanotic infant)by pulse oximeter and lasting >10 seconds. Immediately rescued with rhythmic NC-AC. If the oxygen saturation did not reach to its acceptable level (>85%) within 2 minutes, then traditional CPR procedures involving bag-mask ventilation, ET intubation, Ambu bag ventilation or even chest compressions were substituted.
Mean blood pressure (mmHg) | Participants will continually monitoring by sphygmomanometer for 2 days after the procedure.
  During and after the FB procedure, vital signs are continually monitoring. When the mean blood pressure <50mmHg (measured by continuous non-invasive sphygmomanometer every 5 minutes and one hour, respectively) and lasting morethan one hour. Immediately rescued with rhythmic NC-AC. If the mean BP did not reach to its acceptable level (>50mmHg) within 10 minutes, then traditional CPR procedures involving bag-mask ventilation, ET intubation, Ambu bag ventilation or even chest compressions were substituted.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jue Soong, MD, Principal Investigator — Department of Pediatrics; Taipei-Veteran General Hospital
Locations (1):
- Taipei-Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Soong WJ, Shiao AS, Jeng MJ, Lee YS, Tsao PC, Yang CF, Soong YH. Comparison between rigid and flexible laser supraglottoplasty in the treatment of severe laryngomalacia in infants. Int J Pediatr Otorhinolaryngol. 2011 Jun;75(6):824-9. doi: 10.1016/j.ijporl.2011.03.016. Epub 2011 Apr 21. PMID 21513991